CLINICAL TRIAL: NCT06212011
Title: Investigation on the Effect of Functional Neuromuscular Electrical Stimulation Technique Applied to the Lumbar Multifidus Muscle On Body Kinetics and Kinematics During Sit to Stand Activity In Individuals With Nonspecific Low Back Pain
Brief Title: Effect of Neuromuscular Electrical Stimulation Applied to the Lumbar Multifidus Muscle on Sit to Stand Kinematics in Individuals With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Duygu Yilmaz, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204574
Record Dates: First submitted 2023-12-24; First posted 2024-01-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
Keywords: low back pain; electric stimulation; sit to stand; kinetic; kinematic
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Functional Neuromuscular Electrical Stimulation Group (Experimental): Functional NMES involves stimulating the lumbar multifidus muscle while the individual performs a sit-to-stand activity.
  Interventions: Other: Functional Neuromuscular Electrical Stimulation
- Conventional Neuromuscular Electrical Stimulation Group (Experimental): Conventional NMES intervention involves only stimulating the lumbar multifidus muscle while the individual is in the prone position, and the individual will not reveal any voluntary contraction during stimulation.
  Interventions: Other: Conventional Neuromuscular Electrical Stimulation

INTERVENTIONS:
Other: Functional Neuromuscular Electrical Stimulation — The functional NMES technique involves the application of electrical stimulation during functional activity. In our study, in the functional neuromuscular electrical simulation group, neuromuscular electrical stimulation will be applied to the lumbar multifidus muscle while individuals perform the activity of standing up from sitting.
  Arms: Functional Neuromuscular Electrical Stimulation Group
Other: Conventional Neuromuscular Electrical Stimulation — The conventional neuromuscular electrical simulation technique, electrical stimulation is applied without the individual performing voluntary contractions. In our study, conventional NMES will be applied to the lumbar multifidus muscle with the individual lying in the prone position and the individual will not elicit any voluntary contractions during the simulation.
  Arms: Conventional Neuromuscular Electrical Stimulation Group

SUMMARY:
The goal of this randomized controlled trial, is to investigate the effect of functional NMES and conventional NMES applied to the lumbar multifidus muscle on body kinematic and kinetic values during the sit-to-stand in individuals with non-specific low back pain. Our study will include 24 participants between the ages of 18-65. Which physiotherapy intervention will be applied to the participants will be determined by the block randomization method, using a table of random numbers. After randomization; NMES to the participants' lumbar multifidus muscle during physiotherapy intervention will be applied in two groups; In the first group, NMES will be applied with the conventional technique during prone position and in the second group, NMES will be applied with the functional technique during the sit-to-stand activity. Evaluations will be made twice for each participant- before and after the intervention. During the evaluation, data regarding the change in body kinetics and kinematics of individuals during the sit-to-stand activity will be recorded with a Vicon camera system. For secondary outcome measures, a visual analog scale will be used to evaluate pain, the Roland Morris Disability Questionnaire and the Oswestry Disability Index will be used to evaluate functional status, and the Tampa Kinesiophobia Scale will be used to evaluate fear-avoidance behavior.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic low back pain (12 weeks<)
* Pain in the lumbar and/or hip area (VAS>3)
* Volunteering to participate in the study

Exclusion Criteria:

* History of neurological, metabolic, cardiovascular disease
* Having had spinal surgery, specific lumbar pathology, scoliosis, pregnancy, history of systemic or degenerative disease
* Musculoskeletal system pathology in the last year
* Body mass index being over 30 kg/m2
* Continuing any exercise program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Changes in kinematics of the Lumbar Spine and Hip During sit-to-stand activity | Baseline and first week after 8-week intervention
  With kinematic analysis, the mean, minimum and maximum range of motion of the lumbar spine and hip joint during the sit-to-stand activity will be evaluated and recorded in degrees using the vicon motion capture system (Vicon, 6xVantage 5 Cameras 5MP@420FPS, 2xVue Video Cameras).
Changes in ground reaction force during sit-to-stand activity | Baseline and first week after 8-week intervention
  Ground reaction force will be evaluated using force plates (2xAMTI force plates).

SECONDARY OUTCOMES:
Hip and Lumbar spine range of motion | Baseline and first week after 8-week intervention
  Hip and Lumbar spine range of motion will be evaluated using goniometer and recorded in degrees.
Shortness of the hip flexor, knee flexor and plantar flexor muscles | Baseline and first week after 8-week intervention
  Shortness of the hip flexor, knee flexor and plantar flexor muscles will be evaluated by Thomas test, popliteal angle hamstring test and ankle dorsiflexion ROM measurements, respectively. Results will be recorded in degrees.
Beighton test | Baseline and first week after 8-week intervention
  The Beighton test is a screening technique for hypermobility. The test is a nine-point scale and requires the performance of 5 maneuvers.
Visual analogue scale | Baseline and first week after 8-week intervention
  Visual analog scale will be used to evaluate pain. The visual analog scale consists of a single 10 cm line used to evaluate pain intensity. Patients will be asked to mark the severity of their pain at rest, during activity and during night.
Oswestry Disability Index | Baseline and first week after 8-week intervention
  Oswestry Disability Index will be used to evaluate the degree of loss of function. Higher values represent greater disability.
Roland-Morris Disability Questionnaire | Baseline and first week after 8-week intervention
  Roland-Morris Disability Questionnaire will be used to evaluate functional disabilities. Higher values represent greater disability.
Tampa Kinesiophobia Scale | Baseline and first week after 8-week intervention
  Tampa Kinesiophobia Scale will be used to evaluate fear of movement/reinjury. Higher values represent greater kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)